CLINICAL TRIAL: NCT06790108
Title: Validation of an AI-Assisted Mediastinal EUS System for Training Improvement: a Prospective, Multi-Center, Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: ZhuZhou Central Hospital (Other); The First Affiliated Hospital of University of South China (Other); The First People's Hospital of Chenzhou (Unknown); the Affiliated Nanhua Hospital, University of South China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2023-EUS-AI-002-2
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Mediastinal Disease
MeSH Terms: conditions — Mediastinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-assisted group (Experimental): Endoscopists perform scans with the assistance of AI device.
  Interventions: Device: Artificial intelligence device
- Control group (Placebo Comparator): Endoscopists perform scans without the assistance of AI device.
  Interventions: Device: Artificial intelligence device

INTERVENTIONS:
Device: Artificial intelligence device — This AI device can provide prompts for standard sites of pancreatic scans and anatomical structures. It may also suggest the next operation methods.

SUMMARY:
The goal of this clinical trial is to verify the auxiliary role of the artificial intelligence (AI) system in mediastinal endoscopic ultrasound (EUS) scans. The main questions it aims to answer are as follows:

1. A comparison of the image recognition accuracy between the AI system and EUS endoscopists.
2. Whether the AI system can improve the quality of mediastinal scans for EUS endoscopists.

Participants will conduct mediastinal EUS with or without the assistance of the AI system.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, <80 years old 2.Patients who need endoscopic ultrasonography; 3. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be selected for this trial:

First. The patient's physical condition does not meet the requirements of conventional endoscopic ultrasonography:

Poor physical condition, including hemoglobin ≤8.0g/dl, severe cardiopulmonary insufficiency, etc. Anesthesia assessment failed Pregnancy or breastfeeding In the acute stage of chemical and corrosive injury, it is very easy to cause perforation Recent acute coronary syndrome or clinically unstable ischemic heart attack Heart disease patients with right-to-left shunt, patients with severe pulmonary hypertension (pulmonary artery pressure> 90mmHg), patients with uncontrolled systemic hypertension and patients with adult respiratory distress syndrome.

Second. Disagree to participate in this study.

Third. There are other problems that do not meet the requirements of this research or that affect the results of the research:

1. Mediastinal lesions have previously undergone surgery or radiotherapy and chemotherapy;
2. Mental illness, drug addiction, inability to express themselves or other diseases that may affect follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The completeness for standard station scanning | 1 year
  The primary outcome measure was the completeness for standard station scanning of EUS by endoscopists in the two groups. This was calculated as the number of stations successfully scanned divided by the total number of stations that should have been scanned.

SECONDARY OUTCOMES:
The completeness of anatomical structure scanning | 1 year
  It calculated as the number of anatomical structures successfully scanned divided by the total number of structures that should have been scanned.
Procedure time | 1 year
  It defined as the observation time only, excluding the time spent on puncture, elastography, contrast-enhanced ultrasound, or other lesion observation or treatment.
The incidence of adverse events | 1 year
  The incidence of adverse events in both groups during the entire research process.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, Doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Some data underlying this trial cannot be shared publicly due to protection of participant's privacy.